CLINICAL TRIAL: NCT00817843
Title: Multicenter,Double Blind,Randomized, 2-period, Crossover Study to Compare Ezetimibe/Simvastatin (10mg/10 mg) Combination Tablet Versus Simvastatin 80mg Tablet on Postprandial Arterial Endothelial Function in Patients With Metabolic Syndrome
Brief Title: The PostprAndial eNdothelial Function After Combination of Ezetimibe and simvAstatin Study
Acronym: PANACEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: dr.Frank L.J. Visseren (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, dr.Frank L.J. Visseren, Professor F.L.J. Visseren, MD PhD, head of department of Vascular Medicine, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Vasc-UMCU-10B; 2008-003908-61 (EudraCT Number)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Metabolic Syndrome
Keywords: Postprandial hypertriglyceridemia; Metabolic syndrome; Endothelial function; Flow mediated dilatation; EndoPAT; Simvastatin; Ezetimibe
MeSH Terms: conditions — Metabolic Syndrome | interventions — Simvastatin; Ezetimibe, Simvastatin Drug Combination; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Simva 80mg then Simvai/Eze10/10mg (Experimental): First 6 weeks of Simvastatin 80mg, then 6 weeks of Simvastatin/Ezetimibe 10/10mg after 6 weeks of placebo washout
  Interventions: Drug: Simvastatin; Drug: Simvastatin/Ezetimibe
- First Simva/Eze 10/10mg then Simva 80mg (Experimental): First 6 weeks of Simvastatin/Ezetimibe 10/10mg, then 6 weeks of Simvastatin 80mg after 6 weeks of placebo washout
  Interventions: Drug: Simvastatin; Drug: Simvastatin/Ezetimibe

INTERVENTIONS:
Drug: Simvastatin — 6 weeks of treatment with simvastatin 80 mg
  Other Names: Simvastatin (Zocor)
Drug: Simvastatin/Ezetimibe — 6 weeks of treatment with simvastatin 10 mg / ezetimibe 10 mg combination
  Other Names: Simvastatin/Ezetimibe (Zetia)

SUMMARY:
The purpose of this study is to investigate whether low-dose simvastatin in combination with ezetimibe in comparison to high-dose simvastatin alone, has a beneficial effect on the function of the endothelium after an oral fat load in patients with metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome is defined as a group of cardiovascular risk factors and is mainly driven by the epidemic of obesity. High blood lipid levels after a meal may be an important risk factor for cardiovascular disease. In this study we will investigate whether simvastatin in combination with ezetimibe vs. simvastatin alone, has a beneficial effect on the lipid levels after a meal, but more importantly, whether we can measure a difference in function of the endothelium. In a small pilot study we already found that the combination had a beneficial effect in comparison with simvastatin alone. Now we want to solidify these findings in a larger study.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient has a diagnosis of metabolic syndrome according to the modified 2005 AHA/NHLBI Scientific Statement with at least:

   - Abdominal obesity defined as:

   *Males: waist circumference >102cm
   * Females: waist circumference >88cm and two of the following 4 other criteria:

     - Triglycerides>150 mg/dL

     - HDL Cholesterol
   * Males: HDL-C<40 mg/dL
   * Females:HDL-C<50 mg/dL - Blood pressure
   * Systolic Blood Pressure ≥130 mmHg or
   * Diastolic Blood Pressure ≥85 mmHg

     * Fasting glucose ≥ 100 mg/dL
2. Patient understands the study procedures, alternative treatments available, and risks involved with the study, and voluntarily agrees to participate by giving written informed consent.
3. Patient is a male or female of 18-79 years of age on the day of signing informed consent.
4. Patient is a non-smoker.
5. Patient is willing to maintain a stable diet for the duration of the study.
6. Patient is a postmenopausal female who is not receiving hormone therapy (including cyclic and non-cyclical hormone replacement therapy or any estrogen antagonist/agonist). Postmenopausal status is defined as (1) no menses for ≥1 year but <3 years and confirmed by FSH levels elevated into the postmenopausal range (as defined by the designated laboratory) or (2) no menses for at least 3 years.
7. Patient is naïve to lipid-lowering therapy. Naïve is defined as not being treated with a statin, a fibrate or ezetimibe for 3 months before Visit 1 (Week -2)
8. Patient has a baseline fasting LDL-C level of ≥ 100 mg/dL and < 220 mg/dL, and TG level < 400 mg/dL.

EXCLUSION CRITERIA:

1. Patient has a BMI > 35.
2. Patient has hypersensitivity or intolerance to ezetimibe or simvastatin or any component of these medications, or to latex.
3. Patient routinely consumes more than 14 alcoholic drinks per week.
4. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent.
5. Patient has a smoking history > 10 pack-years (1 pack-year = at least 20 cigarettes per day for a year) OR patient who has smoked within 3 months prior to Visit 1 (Week -2).
6. Patient has exclusionary laboratory values at Visit 1 (Week -2) as listed in the table below:

   liver transaminases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) > 1.5 X ULN with no active liver disease Serum glucose > 7.0 mmol/L Creatine kinase(CK)> 2 X ULN Albumin:creatinine ratio > 34 TSH <0.3 mcIU/mL or > 5.0 mcIU/mL
7. Patient has a history or current evidence of any condition, therapy, lab abnormality or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate.
8. It is not possible to obtain a FMD measurement of sufficient quality at screening (Visit 1)
9. Patient has congestive heart failure, atherosclerotic vascular disease or acute or chronic coronary heart disease.

13. Patient has had a partial ileal bypass, gastric bypass, gastric banding, celiac disease or other significant intestinal malabsorption.

15. Patient has untreated and uncontrolled hypertension with systolic blood pressure >160 mm Hg or diastolic >100 mm Hg at Visit 1 (Week -2). (Patients with untreated hypertension and with office BP at Visit 1 and Visit 2 averaging 160/100 or less can be enrolled). Patients using blood pressure-lowering medication are excluded.

16. Patient has estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 based on the 4-variable MDRD

17. Patient has uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins at Visit 1 (Week -2).

18. Patient has diabetes mellitus defined as a history of diabetes or fasting serum glucose > 126 mg/dL.

For the full exclusion criteria, please check the protocol

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank LJ Visseren, MD PhD, Principal Investigator — UMC Utrecht
Locations (5):
- Netherlands (4):
  - Department of Vascular Medicine UMC Utrecht, Utrecht, Utrecht
  - Academic Medical Center, Amsterdam
  - Vascular Research Center Hoorn, Hoorn
  - Tweesteden Ziekenhuis, Waalwijk
- Hospital Arnau de Vilanova, Lleida, Spain

REFERENCES:
- [Background] Olijhoek JK, Hajer GR, van der Graaf Y, Dallinga-Thie GM, Visseren FL. The effects of low-dose simvastatin and ezetimibe compared to high-dose simvastatin alone on post-fat load endothelial function in patients with metabolic syndrome: a randomized double-blind crossover trial. J Cardiovasc Pharmacol. 2008 Aug;52(2):145-50. doi: 10.1097/FJC.0b013e31817ffe76. PMID 18670365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between and patients were screened of which subjects were randomized in the following centers UMC Utrecht, Utrecht, the Netherlands AMC, Amsterdam, the Netherlands Vascular Research Center, Hoorn, the Netherlands Tweesteden Ziekenhuis, Waalwijk, the Netherlands Hospital Arnau de Vilanova, Lleida, Spain
Pre-assignment Details: Prior to randomization subjects were given a 2 week placebo controled run-in phase to test for adequate compliance.
Groups:
- Simvastatin 80mg First, Then Simvastatin/Ezetimibe 10/10mg: First 6 weeks of treatment with simvastatin 80 mg with placebo, followed by 6 weeks of placebo controlled washout and 6 weeks of simvastatin/ezetimibe 10/10 mg combination and placebo
- Simvastatin/Ezetimibe 10/10mg First, Then Simvastatin 80mg: First 6 weeks of treatment with simvastatin/ezetimibe 10/10 mg combination with placebo, followed by 6 weeks of placebo controlled washout and 6 weeks of simvastatin 80 mg and placebo
Period: First Period (6 Weeks)
Arm/Group | Simvastatin 80mg First, Then Simvastatin/Ezetimibe 10/10mg | Simvastatin/Ezetimibe 10/10mg First, Then Simvastatin 80mg
Started | 50 | 50
Completed | 42 (All patients with >=1 postrandomization dose and measurement were analyzed) | 46
Not Completed | 8 | 4
Period: Washout Period (6 Weeks)
Arm/Group | Simvastatin 80mg First, Then Simvastatin/Ezetimibe 10/10mg | Simvastatin/Ezetimibe 10/10mg First, Then Simvastatin 80mg
Started | 42 | 46
Completed | 41 | 45
Not Completed | 1 | 1
Period: Second Period (6 Weeks)
Arm/Group | Simvastatin 80mg First, Then Simvastatin/Ezetimibe 10/10mg | Simvastatin/Ezetimibe 10/10mg First, Then Simvastatin 80mg
Started | 41 | 45
Completed | 41 (All patients with >=1 postrandomization dose and measurement were analyzed) | 44
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Simvastatin 80mg or Simvastatin/Ezetimibe 10/10mg: All patients were randomized to receive either Simvastatin 80mg or Simvastatin/Ezetimibe 10/10mg during this period
Arm/Group | Simvastatin 80mg or Simvastatin/Ezetimibe 10/10mg
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 60
Region of Enrollment [Number; unit: participants]
  Spain | 16
  Netherlands | 84

OUTCOME MEASURES:

1. Secondary Outcome: Postprandial Endopat Measurement
Time Frame: after 6 weeks of treatment (crossover)
Reporting Status: Not Posted

2. Secondary Outcome: Preprandial Endothelial Function Measured by FMD
Time Frame: after 6 weeks of treatment (crossover)
Reporting Status: Not Posted

3. Secondary Outcome: Preprandial Endopat Measurement
Time Frame: after 6 weeks of treatment (crossover)
Reporting Status: Not Posted

4. Primary Outcome: Treatment Difference in (Postprandial-Fasting) FMD
Description: A comparison of the postprandial minus fasting change in FMD under treatment with simvastatin 80 mg versus simvastatin 10/10 mg
Time Frame: After 6 weeks of treatment
Population: Analyses were performed in randomized patients who received ≥1 dose of study treatment and who had a post-randomization analysis measurement
Measure: Mean (Standard Error); unit: % (change FMD)
Groups:
- Simvastatin 80 mg: 6 weeks of treatment with simvastatin 80 mg
- Simvastatin 10 mg / Ezetimibe 10 mg: 6 weeks of treatment with simvastatin 10 mg / ezetimibe 10 mg
Arm/Group | Simvastatin 80 mg | Simvastatin 10 mg / Ezetimibe 10 mg
Number analyzed (Participants) | 91 | 90
% (change FMD) | -0.34 (0.210) | -0.43 (0.202)
Statistical Analysis 1: Comparison: Simvastatin 80 mg vs Simvastatin 10 mg / Ezetimibe 10 mg; Between treatment difference in the change in FMD from the fasting to the post-fat load state. Null hypothesis was that combination therapy (simvastatin/ezetimibe) would protect the FMD in the post-fat load phase and would therefore be associated with a smaller drop in FMD Power calculation was based on the results from a pilot study. To detect a 1.0% difference between treatments with a SD of 2.7% and a power of 90% (alfa 0.05, two tailed) 80 evaluable patients were needed; Test type: Superiority or Other; p = 0.766, ANOVA; Mean Difference (Final Values) = -0.09, Standard Error of Mean 0.295

ADVERSE EVENTS:
Arm/Group | Simvastatin 80mg or Simvastatin/Ezetimibe 10/10mg
Serious Adverse Events (participants affected / at risk) | 2/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin 80mg or Simvastatin/Ezetimibe 10/10mg (N=100)
Myocardial infarction (Vascular disorders) | 1 (1) — During placebo washout
Appendicitis (Gastrointestinal disorders) | 1 (1) — During placebo washout phase

LIMITATIONS AND CAVEATS:
One limitation is that the study was conducted in obese patients with the metabolic syndrome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No